CLINICAL TRIAL: NCT00339105
Title: The Usefulness of HyperQ Recordings for the Early Diagnosis of Acute Coronary Syndrome in Patients Presenting With Chest Pain
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Other Study IDs: SHEBA-06-4114-SM-CTIL
Record Dates: First submitted 2006-06-19; First posted 2006-06-20 (Estimated); Last update posted 2007-01-17 (Estimated); Status verified 2007-01

CONDITIONS: Acute Coronary Syndrome
Keywords: Acute; Coronary; Syndrome; HyperQ; High; Frequency; ECG; chest; pain
MeSH Terms: conditions — Acute Coronary Syndrome; Syndrome; Pain

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
The purpose of the study is to assess the usefulness of high Frequency mid-QRS analysis in identifying the ischemic origin of patients presenting to the Emergency Room (ER)with Chest pain.

DETAILED DESCRIPTION:
Introduction:

Chest pain is the leading cause of urgent admission to the Emergency Department (ED) in western countries.Acute Coronary Syndrome(ACS) continues to be among the most difficult to predict or diagnose. Misdiagnoses may lead to discharge of patients with ACS, who should have been admitted as well as costly unnecessary hospitalizations of patients who do not have ACS.

Objectives:

To evaluate the usefulness of High Frequency mid-QRS analysis in identifying the ischemic patients out of all patients presenting to the Emergency Room (ER) with chest pain.

Comparisons:

A continuous High Frequency Mid-QRS recording will be performed using the HyperQ System (BSP Ltd.) and compared to clinical, electrophysiologic and laboratory results. The golden standards used to compare the methods will be either CT-Angio, Echocardiography or Cardiac SPECT. A follow-up inquiry will be performed after 3 months and Coronary Angiography results will be sought and compared as well.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Patients with chest pain, with possible ACS.
* Patients admitted to the 'chest pain unit'
* Chest pain appeared within 24 hours prior to admission to the 'chest pain unit'
* No history of trauma or any other evident medical cause of chest pain
* Signed an Informed Consent

Exclusion Criteria:

* Implanted pacemaker or defibrillator
* History of trauma or other evident medical cause of chest pain
* Patients admitted to Intensive Cardiac Care Unit or intermediate Cardiac Care Unit
* Patients discharged from the ER
* Patients with Bundle-Branch-Block or other intra-ventricular delay of more than 120 mSec

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2006-06; Study Completion 2007-01

CONTACTS AND LOCATIONS:
Overall Officials: Shlomi Matetzky, MD, Principal Investigator — Head of Chest Pain Unit, ER, Sheba Medical Center
Locations (1):
- The Chest Pain Unit, ER, Sheba Medical Center, Tel-Hashomer, Ramat Gan, Israel

REFERENCES:
- [Background] Abboud S, Zlochiver S. High-frequency QRS electrocardiogram for diagnosing and monitoring ischemic heart disease. J Electrocardiol. 2006 Jan;39(1):82-6. doi: 10.1016/j.jelectrocard.2005.09.007. No abstract available. PMID 16387057
- See also: BSP Ltd. is the company that developed the HyperQ system — http://www.bsp.co.il